CLINICAL TRIAL: NCT02258971
Title: Investigation of the Metabolism and Pharmacokinetics of 1200 μg (Free Cation) [14C] BEA 2180 BR Administered Orally Compared to 500 μg (Free Cation) [14C] BEA 2180 BR Administered Intravenously in Healthy Male Volunteers in an Open Label, Single-dose and Parallel Study Design
Brief Title: Metabolism and Pharmacokinetics of [14C] BEA 2180 BR Administered Orally Compared to [14C] BEA 2180 BR Administered Intravenously in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1205.8
Record Dates: First submitted 2014-10-01; First posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (2):
- BEA 2180 BR oral (Experimental)
  Interventions: Drug: BEA 2180 BR oral
- BEA 2180 BR infusion (Active Comparator)
  Interventions: Drug: BEA 2180 BR infusion

INTERVENTIONS:
Drug: BEA 2180 BR oral — Oral solution
  Arms: BEA 2180 BR oral
Drug: BEA 2180 BR infusion — Solution for infusion to be reconstituted with isotonic saline
  Arms: BEA 2180 BR infusion

SUMMARY:
Primary objectives: To determine the basic pharmacokinetics of BEA 2180 BR, its metabolites CD 1975 ZW and CD 1976 ZW and radioactivity including excretion mass balance, excretion pathways and metabolism following the oral and intravenous administration of [14C] BEA 2180 BR

Secondary objectives: To determine safety and tolerability following single dose oral and iv administration of BEA 2180 BR in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age ≥35 and Age ≤70 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Subjects must agree to minimize the risk of female partners becoming pregnant from the dosing day until 3 months after the completion of the study. Acceptable methods of contraception for male volunteers include a vasectomy no less than 3 months prior to dosing, barrier contraception or a medically accepted contraceptive method. For female partners of male volunteers, acceptable methods of contraception include intra-uterine device, tubal ligation, hormonal contraceptive since at least two months and diaphragm with spermicide
5. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including blood pressure (BP), pulse rate (PR) and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to study drug or its excipients)
8. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within two months prior to administration or during the trial
11. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
12. Inability to refrain from smoking during the stay in the trial centre
13. Alcohol abuse (more than 2 units of alcoholic beverages per day or more than 14 units per week (1 unit equals 1 pint [285 mL] of beer or lager, 1 glass [125 mL] of wine, 25 mL shot of 40% spirit)more than 60 g/day).
14. Drug abuse
15. Blood donation (more than 100 mL within 60 days prior to study drug administration or during the trial)
16. Excessive physical activities (within one week prior to administration or during the trial until follow-up examination)
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of study centre
19. A marked baseline prolongation of QT/Heart rate-corrected QT interval (QTc) interval (e.g., repeated demonstration of a QTc interval >450 ms)

    Exclusion criteria specific for this study:
20. Veins unsuitable for infusion and blood sampling
21. Pulse rate (PR) interval >220 ms or QRS interval >120 ms
22. Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column)), during work or during participation in a medical trial in the previous year
23. Irregular defecation pattern (less than once per 2 days)

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Individual time course profiles of [14C] radioactivity | Up to 312 hours after drug administration
Individual time course profiles of BEA 2180 and its metabolites CD 1975 ZW and CD 1976 ZW | Up to 312 hours after drug administration
Rate and extent of excretion mass balance based on the total radioactivity in urine and faeces | Up to 312 hours after drug administration
Elucidation of metabolite structures and identification of major metabolites in plasma, urine, and faeces (if feasible) in comparison with various animal species | Up to 312 hours after drug administration
Cblood cells/Cplasma ratio of [14C] -radioactivity | Up to 96 hours after drug administration
Cmax (maximum concentration of the analyte(s) in plasma) | Up to 96 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte(s) in plasma) | Up to 96 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte(s) in plasma over the time interval from 0 to the time of the last quantifiable data point) | Up to 96 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte(s) in plasma over the time interval from 0 to infinity) | Up to 96 hours after drug administration
λz (terminal rate constant in plasma) | Up to 96 hours after drug administration
t1/2 (terminal half-life of the analyte(s) in plasma) | Up to 96 hours after drug administration
MRT (mean residence time of the analyte(s) in the body) | Up to 96 hours after drug administration
CL (total clearance of the analyte in plasma) | Up to 96 hours after drug administration
Vz (apparent volume of distribution during the terminal phase λz) | Up to 96 hours after drug administration
Vss (apparent volume of distribution at steady state) | Up to 96 hours after drug administration
fe0-tz (amount of analyte excreted in urine within the time interval zero to tz in % of dose) | Up to 312 hours after drug administration
fefaeces,0-tz (amount of analyte excreted in faeces within the time interval zero to tz in %) of dose, additionally excretion within each sampling interval will be calculated) | Up to 312 hours after drug administration
CLR,0-tz (renal clearance of analyte) | Up to 96 hours after drug administration
Fa (fraction of drug absorbed after oral administration based on radioactivity data) based on oral and i.v. data | Up to 96 hours after drug administration

SECONDARY OUTCOMES:
Number of participants with abnormal findings in physical examination | Up to day 29 after first drug administration
Number of participants with clinically significant changes in vital signs | Up to day 29 after first drug administration
Number of participants with abnormal findings in 12-lead ECG | Up to day 29 after first drug administration
Number of participants with abnormal changes in clinical laboratory parameters | Up to day 29 after first drug administration
Number of participants with adverse events | Up to day 29 after first drug administration
Investigator global clinical assessment on a 4-point scale | Up to day 15 after first drug administration
Investigator assessed local tolerability on a 6-point scale | Up to day 15 after first drug administration